CLINICAL TRIAL: NCT03233230
Title: A Phase IIb, Randomized, Double-blind Study in Subjects With Rheumatoid Arthritis Evaluating the Safety and Efficacy of Evobrutinib Compared With Placebo in Subjects With an Inadequate Response to Methotrexate
Brief Title: Phase IIb Study of Evobrutinib in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS200527-0060; 2017-000384-32 (EudraCT Number)
Record Dates: First submitted 2017-07-25; First posted 2017-07-28 (Actual); Results first posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; American College of Rheumatology; High-sensitivity C-reactive protein; Bruton's tyrosine kinase
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — evobrutinib; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- M2951 25 mg QD (Experimental)
  Interventions: Drug: M2591 25 mg QD
- M2951 75 mg QD (Experimental)
  Interventions: Drug: M2951 75 mg QD
- M2951 50 mg BID (Experimental)
  Interventions: Drug: M2951 50 mg BID

INTERVENTIONS:
Drug: M2591 25 mg QD — Participants received 25 milligrams (mg) of M2951 orally once daily (QD) for 12 weeks.
  Other Names: Evobrutinib
  Arms: M2951 25 mg QD
Drug: M2951 75 mg QD — Participants received 75 mg of M2951 orally QD for 12 weeks.
  Other Names: Evobrutinib
  Arms: M2951 75 mg QD
Drug: M2951 50 mg BID — Participants received 50 mg of M2951 orally twice daily (BID) for 12 weeks.
  Other Names: Evobrutinib
  Arms: M2951 50 mg BID
Drug: Placebo — Participants received placebo matched to M2951 orally for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine the efficacy, dose response, and safety of M52951 in participants with Rheumatoid Arthritis (RA), and to consider a dose to took forward into Phase III development.

ELIGIBILITY:
Inclusion Criteria:

* In Japan, if a participant is less than (<) 20 years, the written informed consent from the participant's parent or guardian will be required in addition to the participant's written consent.
* Confirmed diagnosis of RA according to 2010 ACR/EULAR RA classification criteria of at least 6 months duration prior to Screening
* Persistently active moderate to severe RA at both Screening and Randomization (if significant surgical treatment of a joint has been performed, that joint cannot be counted for entry or enrollment purposes), as defined by: >= 6 swollen joints (of 66 assessed) and >= 6 tender joints (of 68 assessed).
* An hsCRP >= 5.0 milligram/liter (mg/L) at Screening
* Treatment for >= 16 weeks with 7.5 to 25 mg/week Methotrexate (MTX) at a stable dose and route of administration (oral or parenteral) for at least 8 weeks prior to dosing with the Investigational Medicinal Product (IMP) and maintained throughout the trial
* For participants entering the trial on MTX doses < 15 mg/week (< 10 mg/week in Japan), there must be clear documentation in the medical record that higher doses of MTX were not tolerated or that the dose of MTX is the highest acceptable dose based on local clinical practice guidelines.
* For MRI Sub-study participants, participants must have palpable synovitis of the wrist and/or >= 1 of metacarpophalangeal joints 1 to 5, defined as loss of bony contours with palpable joint effusion and/or swelling, in the MRI-designated hand (that is., the hand being used in MRI assessments).

Exclusion Criteria:

* ACR functional class IV as defined by the ACR classification of functional status or wheelchair/bedbound
* Use of oral corticosteroids greater than (>) 10 mg daily prednisone equivalent, or change in dose of corticosteroids within 2 weeks prior to Screening or during Screening
* Use of injectable corticosteroids (including intra-articular corticosteroids) or intra-articular hyaluronic acid within 4 weeks prior to Screening or during Screening
* Initiation or change in dose for nonsteroidal anti-inflammatory drugs (NSAIDs) (including low-dose aspirin and cyclooxygenase-2 inhibitors) within 2 weeks prior to dosing with the IMP
* High potency opioid analgesics are prohibited within 2 weeks prior to Screening and during the trial; other analgesics are allowed (that is, acetaminophen, codeine, hydrocodone*, propoxyphene*, or tramadol), although not within 24 hours of study visits with clinical assessments (*not approved in Japan)
* Current or prior treatment with any of the following:
* Biologic Disease-modifying anti-rheumatic drugs (DMARDs) (approved or investigational), including but not limited to:
* Tumor necrosis factor (TNF) antagonists or biosimilars of these agents (approved or investigational), or any investigational TNF antagonist
* Interleukin-6 antagonists
* Abatacept (CTLA4-Fc)
* Anakinra* (IL-1 receptor antagonist) (*not approved in Japan)
* B cell-depleting antibodies (example, rituximab, ocrelizumab*, ofatumumab, obinutuzumab*, ocaratuzumab*, veltuzumab*, or any biosimilars of these agents [approved or investigational]) (*not approved in Japan)
* Anti-BLyS (B lymphocyte stimulator) agents (example, belimumab, tabalumab*) (*not approved in Japan)
* Dual BLyS/A proliferation-inducing ligand (APRIL) neutralizing agents (that is, atacicept*, RCT-18*) (*not approved in Japan)
* Targeted synthetic DMARDs, specifically:
* Janus kinase inhibitors
* Other Bruton's tyrosine kinase (BTK) inhibitors
* Alkylating agents (example, chlorambucil*, cyclophosphamide) (*not approved in Japan).
* The following restrictions on nonbiologic DMARD must be followed:
* Auranofin (Ridaura), minocycline, penicillamine, sulfasalazine, cyclosporine, mycophenolate (mycophenolate sodium not approved in Japan), tacrolimus, azathioprine: must have been discontinued for 4 weeks prior to dosing with the IMP
* Leflunomide (Arava) must have been discontinued 12 weeks prior to dosing with the IMP if no elimination procedure is followed. Alternately, it should have been discontinued with the following elimination procedure at least 4 weeks prior to dosing with the IMP:
* Cholestyramine at a dosage of 8 gram 3 times a day for at least 24 hours, or activated charcoal at a dosage of 50 gram 4 times a day for at least 24 hours.
* Injectable Gold (aurothioglucose* or aurothiomalate): must have been discontinued for 8 weeks prior to dosing with the IMP (*not approved in Japan)
* Anti-malarials (hydroxychloroquine, chloroquine*) will be allowed in this trial. Participants may be taking oral hydroxychloroquine (=< 400 mg/day) or chloroquine (=< 250 mg/day), doses must have been stable for at least 12 weeks prior to dosing with the IMP, and will need to be continued at that stable dose for the duration of the trial. If discontinued prior to this trial, they must have been discontinued for 4 weeks prior to dosing with the IMP (*not approved in Japan).
* For MRI Substudy:
* Inability to comply with MRI scanning, including contraindications to MRI such as known allergy to gadolinium contrast media, claustrophobia (if the site does not have ability to scan extremities only), presence of a pacemaker, cochlear implants, ferromagnetic devices or clips, intracranial vascular clips, insulin pumps, and nerve stimulators.
* More than 25% of applicable joints of the target hand and wrist having had prior surgery or showing maximum Genant-modified Sharp erosion (3.0) or joint-space narrowing (4.0) scores, based on single posteroanterior radiographs of target hand and wrist read centrally.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc.
Locations (98):
- United States (8):
  - Arizona Arthritis & Rheumatology Associates, P.C., Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Phoenix, Arizona
  - East Bay Rheumatology Medical Group, Inc., San Leandro, California
  - Omega Research Consultants, DeBary, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - McIlwain Medical Group, PA, Tampa, Florida
  - Medication Management, LLC, Greensboro, North Carolina
  - Arthritis Clinic Of Central Texas, San Marcos, Texas
- Argentina (13):
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas, Mar del Plata, Buenos Aires
  - Instituto Medico CER, Quilmes, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes, Buenos Aires
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, San Miguel de Tucuman
  - Centro de Investigaciones Reumatológicas, San Miguel de Tucumán, Tucumán Province
  - Organizacion Medica de Investigacion (OMI), Ciudad Autonoma Buenos Aires
  - APRILLUS, Ciudad Autonoma Buenos Aires
  - Expertia S.A- Mautalen Salud e Investigación, Ciudad Autonoma Buenos Aires
  - Hospital General de Agudos Dr. J. M. Ramos Mejia, Ciudad Autonoma Buenos Aires
  - ILAIM-CEOM Inst. Latinoamericano de Inv. Medicas, Córdoba
  - Instituto Reumatológico Strusberg, Córdoba
  - Centro Polivalente de Asistencia e Inv. Clinica CER, San Juan
- Bulgaria (3):
  - MHAT "Hadzhi Dimitar", OOD, Sliven
  - DCC "Alexandrovska", EOOD, Sofia
  - UMHAT "SofiaMed", OOD, Sofia
- Chile (4):
  - Centro Medico Prosalud, Santiago
  - Interin, Santiago
  - BioMedica Research Group, Santiago
  - Centro de Estudios Reumatologicos, Santiago
- Colombia (6):
  - Centro de Reumatologia y Ortopedia SAS, Barranquilla
  - Riesgo de Fractura S.A., Bogotá
  - Simedics Ips Sas, Bogotá
  - Centro de Investigacion en Reumatologia y Especialidades Medicas SAS. CIREEM, Bogotá
  - Servimed S.A.S., Bucaramanga
  - Clinica de Artritis Temprana S.A., Cali
- Czechia (9):
  - Revmatolog, s.r.o, Jihlava
  - CCBR Ostrava s.r.o., Ostrava
  - ARTROSCAN s.r.o., Ostrava - Trebovice
  - CLINTRIAL s.r.o., Prague
  - MUDR. Zuzana URBANOVA Revmatologie, Prague
  - Thomayerova nemocnice, Praha 4 - Krc
  - MUDR. Zuzana URBANOVA Revmatologie, Praha 4 Nusle
  - MEDICAL PLUS s.r.o., Uherské Hradiště
  - PV-MEDICAL s.r.o., Zlín
- Mexico (5):
  - Centro Investigacion en Artritis y Osteoporosis S.C., Mexicali, Baja California Norte
  - Clinica de Investigacion en Reumatologia y Obesidad S.C., Guadalajara, Jalisco
  - RM Pharma Specialists SA de CV, Mexico City, Mexico City
  - Investigacion y Biomedicina de Chihuahua, S.C., Chihuahua City
  - Centro de Investigacion y Atencion Integral Durango CIAID, Durango
- Poland (16):
  - ClinicMed Daniluk, Nowak Spółka Jawna, Bialystok
  - Centrum Reumatologiczne Indywidualna Specjalistyczna Praktyka Lekarska lek. Barbara Bazela, Elblag
  - MCBK Iwona Czajkowska Anna Podrażka- Szczepaniak S.C., Grodzisk Mazowiecki
  - Care Clinic, Katowice
  - Silmedic sp. z o.o, Katowice
  - Indywidualna Specjalistyczna Praktyka Lekarska Maciej Zymla, Knurów
  - Malopolskie Centrum Medyczne s.c., Krakow
  - Grazyna Pulka Specjalistyczny Osrodek "ALL-MED", Krakow
  - GLOBE CLINICAL RESEARCH (Globe Badania Kliniczne Sp z o.o.), Kłodzko
  - Centrum Badan Klinicznych S.C., Poznan
  - RCMed, Sochaczew
  - Medycyna Kliniczna, Warsaw
  - Rheuma Medicus Zaklad Opieki Zdrowotnej, Warsaw
  - Centrum Medyczne AMED, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
  - Reum-Medica S.C Eliza Roszkowska, Wroclaw
- Russia (8):
  - Research Institute of Emergency Medical Care, Saint Petersburg, Sankt-Peterburg
  - Limited Liability Company "Centre of Medical Common Practice", Novosibirsk
  - Ultramed, Omsk
  - SPb SBIH "Clinical Rheumatological Hospital # 25", Saint Petersburg
  - LLC Medical Sanitary Unit#157, Saint Petersburg
  - NIH "Departmental Hospital on Station Smolensk of OJSC "Russian Railways", Smolensk
  - SAIH of Yaroslavl region "Clinical Hospital of Emergency Medical Care n.a. N. V. Solovyev", Yaroslavl
  - SBHI of Yaroslavl Region "Clinical Hospital # 8", Yaroslavl
- Serbia (5):
  - Institute of Rheumatology_Site 1, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Bezanijska kosa, Belgrade
  - Institute of Treatment and Rehabilitation "Niska Banja", Niška Banja
  - General Hospital "Dr Laza K. Lazarevic" Sabac, Šabac
- South Africa (7):
  - Wits Clinical Research, Johannesburg, Gauteng
  - Clinresco Centres (Pty) Ltd, Kempton Park, Gauteng
  - Emmed Research, Pretoria, Gauteng
  - University of Pretoria Clinical Research Unit, Pretoria, Gauteng
  - Naidoo, A, Durban, KwaZulu-Natal
  - Arthritis Clinical Research Trial Unit, Cape Town, Western Cape
  - Winelands Medical Research Centre, Stellenbosch, Western Cape
- Ukraine (14):
  - Regional CH Dep of Rheumatology SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - GI L.T.Malaya Therapy National Institute of the NAMS of Ukraine, Kharkiv
  - Communal Institution of Healthcare Kharkiv City Clinical Hospital #8, Kharkiv
  - Medical Center Medical Clinic Blagomed LLC, Kyiv
  - Med Center 'Ok!Clinic+' of International Institute of Clinical Trials LLC, Kyiv
  - Medical Center of Revmotsentr LLC, Kyiv
  - SI D.F.Chebotariov Institute of Gerontology of NAMSU, Kyiv
  - CH of State Border Service of Ukraine (Military Base 2522) Dept of Therapy, D.Halytskyi Lviv NMU, Lviv
  - M.V. Sklifosovskyi Poltava RCH Dept of Rheumatology HSEIU UMSA, Poltava
  - A.Novak Transcarpathian Regional Clinical Hospital, Uzhhorod
  - National Pirogov Memorial Medical University, Vinnytsia
  - CI City Hospital #1, Zaporizhzhia
  - CI Zaporizhzhia Regional Clinical Hospital of ZRC, Zaporizhzhia
  - CI Zaporizhzhia Regional Clinical Hospital of ZRC, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, EMD Serono will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.emdgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- [Derived] Montalban X, Wallace D, Genovese MC, Tomic D, Parsons-Rich D, Bolay CL, Kao AH, Guehring H. A plain language summary of what clinical studies can tell us about the safety of evobrutinib - a potential treatment for multiple sclerosis. Neurodegener Dis Manag. 2023 Aug;13(4):207-213. doi: 10.2217/nmt-2023-0003. Epub 2023 Jun 22. PMID 37345645
- [Derived] Montalban X, Wallace D, Genovese MC, Tomic D, Parsons-Rich D, Le Bolay C, Kao AH, Guehring H. Characterisation of the safety profile of evobrutinib in over 1000 patients from phase II clinical trials in multiple sclerosis, rheumatoid arthritis and systemic lupus erythematosus: an integrated safety analysis. J Neurol Neurosurg Psychiatry. 2023 Jan;94(1):1-9. doi: 10.1136/jnnp-2022-328799. Epub 2022 Nov 23. PMID 36418156
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200527-0060
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 933 participants with rheumatoid arthritis were screened. Out of which, 390 participants were randomized in ratio of 1:1:1:1 to 1 of the 4 treatment groups: Placebo; M2951 25 milligrams (mg) once daily (QD), M2951 75 mg QD and M2951 50 mg twice daily (BID).
Groups:
- M2951 25 mg QD: Participants received 25 milligrams (mg) of M2951 orally once daily (QD) for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Started | 97 | 98 | 96 | 99
Completed | 82 | 83 | 84 | 91
Not Completed | 15 | 15 | 12 | 8
Not completed — Adverse Event | 6 | 3 | 6 | 3
Not completed — Protocol Violation | 1 | 2 | 1 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Other | 5 | 5 | 5 | 3
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (mITT) analysis set included all randomized participants who received at least one dose of Investigational Medicinal Product (IMP) (M2951 or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID | Total
Number analyzed (Participants) | 97 | 98 | 96 | 99 | 390
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (12.24) | 50.9 (13.15) | 53.3 (11.33) | 53.7 (12.13) | 52.7 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 82 | 76 | 77 | 312
  Male | 20 | 16 | 20 | 22 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 33 | 35 | 38 | 138
  Not Hispanic or Latino | 65 | 65 | 61 | 61 | 252
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 0 | 3
  White | 92 | 94 | 91 | 97 | 374
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved American College of Rheumatology 20 Percent (%) Response Criteria (ACR20) Assessed Using High-Sensitivity C-reactive Protein (hsCRP) at Week 12
Description: ACR20 response: a participant has at least 20% improvement in both tender joint counts (based on a total of 68 joints) and swollen joint counts (based on a total of 66 joints) together with 20% improvement in at least 3 of the following: 1) participant's assessment of pain; 2) participant's global assessment of disease activity; 3) physician's global assessment of disease activity; 4) participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI); and 5) acute phase reactant as measured by high-sensitivity C-reactive protein (hsCRP). Percentage of participants with ACR20 response using hsCRP = Number of participants with ACR20 response using hsCRP divided by total modified intent-to-treat (mITT) participants * 100.
Time Frame: Week 12
Population: The mITT analysis set included all randomized participants who received at least one dose of Investigational Medicinal Product (IMP) (M2951 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 97 | 98 | 96 | 99
percentage of participants | 49.5 | 59.2 | 51.0 | 59.6
Statistical Analysis 1: Comparison: Placebo vs M2951 25 mg QD; Test type: Superiority; p = 0.1746, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.84 to 2.61]
Statistical Analysis 2: Comparison: Placebo vs M2951 75 mg QD; Test type: Superiority; p = 0.8283, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.61 to 1.87]
Statistical Analysis 3: Comparison: Placebo vs M2951 50 mg BID; Test type: Superiority; p = 0.1298, Regression, Logistic; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.88 to 2.74]

2. Secondary Outcome: Percentage of Participants With Low Disease Activity Score (DAS28 Less Than [<] 3.2) Based on 28 Joint Count-High-Sensitivity C-reactive Protein (DAS28-hsCRP) at Week 12
Description: Disease Activity Score (DAS) based on a 28 joint count hsCRP consisted of composite numerical score of following variables: tender joint count (TJC28), swollen joint count (SJC28), hsCRP (mg/mL), and participant's global assessment of disease activity. DAS28-hsCRP was calculated using following formula: DAS28-hsCRP equals to (=) 0.56*square root (sqrt) (TJC28) plus (+) 0.28*sqrt (SJC28) + 0.36*natural log(hsCRP+1) + 0.014* participant's global assessment of disease activity + 0.96. Scores ranged 0-9.4, where lower scores indicated less disease activity. Percentage of participants with low DAS28 < 3.2 based on DAS28- hsCRP at Week 12 were reported.
Time Frame: Week 12
Population: The mITT analysis set included all randomized participants who received at least one dose of IMP (M2951 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 97 | 98 | 96 | 99
percentage of participants | 7.2 | 20.4 | 24.0 | 20.2
Statistical Analysis 1: Comparison: Placebo vs M2951 25 mg QD; Test type: Superiority; p = 0.0077, Cochran-Mantel-Haenszel; Response rate difference = 0.13, 95% CI 2-sided [0.04 to 0.23]
Statistical Analysis 2: Comparison: Placebo vs M2951 75 mg QD; Test type: Superiority; p = 0.0013, Cochran-Mantel-Haenszel; Response rate difference = 0.17, 95% CI 2-sided [0.07 to 0.27]
Statistical Analysis 3: Comparison: Placebo vs M2951 50 mg BID; Test type: Superiority; p = 0.0080, Cochran-Mantel-Haenszel; Response rate difference = 0.13, 95% CI 2-sided [0.04 to 0.23]

3. Secondary Outcome: Percentage of Participants With Remission Disease Activity Score (DAS28 Less Than [<] 2.6) Based on a 28 Joint Count-High-Sensitivity C-reactive Protein (DAS28-hsCRP) at Week 12
Description: Disease Activity Score (DAS) based on a 28 joint count hsCRP consisted of composite numerical score of following variables: tender joint count (TJC28), swollen joint count (SJC28), hsCRP (mg/mL), and participant's global assessment of disease activity. DAS28-hsCRP was calculated using following formula: DAS28-hsCRP equals to (=) 0.56*square root (sqrt) (TJC28) plus (+) 0.28*sqrt (SJC28) + 0.36*natural log(hsCRP+1) + 0.014* participant's global assessment of disease activity + 0.96. Scores ranged 0-9.4, where lower scores indicated less disease activity. A DAS28 score less than (<) 2.6 indicated clinical remission. Percentage of participants with low DAS28 < 2.6 based on DAS28- hsCRP at Week 12 were reported.
Time Frame: Week 12
Population: The mITT analysis set included all randomized participants who received at least one dose of IMP (M2951 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 97 | 98 | 96 | 99
percentage of participants | 1.0 | 10.2 | 10.4 | 10.1
Statistical Analysis 1: Comparison: Placebo vs M2951 25 mg QD; Test type: Superiority; p = 0.0056, Cochran-Mantel-Haenszel; Response rate difference = 0.09, 95% CI 2-sided [0.03 to 0.17]
Statistical Analysis 2: Comparison: Placebo vs M2951 75 mg QD; Test type: Superiority; p = 0.0050, Cochran-Mantel-Haenszel; Response rate difference = 0.09, 95% CI 2-sided [0.03 to 0.17]
Statistical Analysis 3: Comparison: Placebo vs M2951 50 mg BID; Test type: Superiority; p = 0.0053, Cochran-Mantel-Haenszel; Response rate difference = 0.09, 95% CI 2-sided [0.03 to 0.17]

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% Response Criteria (ACR50)
Description: ACR50 response: a participant has at least 50% improvement in both tender joint counts (based on a total of 68 joints) and swollen joint counts (based on a total of 66 joints) together with 50% improvement in at least 3 of the following: 1) participant's assessment of pain; 2) participant's global assessment of disease activity; 3) physician's global assessment of disease activity; 4) participant's assessment of physical function measured by Health Assessment Questionnaire - Disability Index [HAQ-DI]; and 5) acute phase reactant as measured by High-sensitivity C-reactive protein [hsCRP]. Percentage of participants with ACR50 response = Number of participants with ACR50 response divided by total mITT participants * 100.
Time Frame: Week 12
Population: The mITT analysis set included all randomized participants who received at least one dose of IMP (M2951 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 97 | 98 | 96 | 99
percentage of participants | 19.6 | 28.6 | 27.1 | 26.3
Statistical Analysis 1: Comparison: Placebo vs M2951 25 mg QD; Test type: Superiority; p = 0.1419, Cochran-Mantel-Haenszel; Response rate difference = 0.09, 95% CI 2-sided [-0.03 to 0.21]
Statistical Analysis 2: Comparison: Placebo vs M2951 75 mg QD; Test type: Superiority; p = 0.2202, Cochran-Mantel-Haenszel; Response rate difference = 0.07, 95% CI 2-sided [-0.05 to 0.19]
Statistical Analysis 3: Comparison: Placebo vs M2951 50 mg BID; Test type: Superiority; p = 0.2328, Cochran-Mantel-Haenszel; Response rate difference = 0.07, 95% CI 2-sided [-0.05 to 0.19]

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% Response Criteria (ACR70)
Description: ACR70 response: a participant has at least 70% improvement ACR70 response in both tender joint counts (based on a total of 68 joints) and swollen joint counts (based on a total of 66 joints) together with 70% improvement in at least 3 of the following: 1) participant's assessment of pain; 2) participant's global assessment of disease activity; 3) physician's global assessment of disease activity; 4) participant's assessment of physical function measured by Health Assessment Questionnaire - Disability Index [HAQ-DI]; and 5) acute phase reactant as measured by High-sensitivity C-reactive protein [hsCRP]. Percentage of participants with ACR70 response = Number of participants with ACR70 response divided by total mITT participants * 100.
Time Frame: Week 12
Population: The mITT analysis set included all randomized participants who received at least one dose of IMP (M2951 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 97 | 98 | 96 | 99
percentage of participants | 5.2 | 11.2 | 10.4 | 10.1
Statistical Analysis 1: Comparison: Placebo vs M2951 25 mg QD; Test type: Superiority; p = 0.1232, Cochran-Mantel-Haenszel; Response rate difference = 0.06, 95% CI 2-sided [-0.02 to 0.15]
Statistical Analysis 2: Comparison: Placebo vs M2951 75 mg QD; Test type: Superiority; p = 0.1725, Cochran-Mantel-Haenszel; Response rate difference = 0.05, 95% CI 2-sided [-0.03 to 0.14]
Statistical Analysis 3: Comparison: Placebo vs M2951 50 mg BID; Test type: Superiority; p = 0.1795, Cochran-Mantel-Haenszel; Response rate difference = 0.05, 95% CI 2-sided [-0.03 to 0.13]

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs According to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 4.03 (NCI-CTCAE v4.03)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a participant, which does not necessarily have causal relationship with treatment. A serious AE was defined as an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inparticipant hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs: events between first dose of study drug that were absent before treatment/that worsened relative to pre-treatment state up to 16 weeks. TEAEs included both serious TEAEs and non-serious TEAEs. Number of participants with TEAEs and serious TEAEs were reported.
Time Frame: up to Week 16
Population: The safety analysis set (SAF) included all participants who received at least 1 dose of IMP (M2951 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 97 | 98 | 96 | 99
Participants
  TEAEs | 44 | 48 | 48 | 50
  Serious TEAEs | 2 | 2 | 2 | 1

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Severity According to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 4.03 (NCI-CTCAE v4.03)
Description: Severity of TEAEs were graded using NCI-CTCAE v4.03 toxicity grades, as follows: Grade 1= Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life-threatening and Grade 5 = Death. Number of participants with TEAEs by severity were reported.
Time Frame: up to Week 16
Population: The SAF included all participants who received at least 1 dose of IMP (M2951 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 97 | 98 | 96 | 99
Participants
  Grade 1 | 33 | 42 | 37 | 40
  Grade 2 | 19 | 14 | 23 | 17
  Grade 3 | 2 | 5 | 1 | 1
  Grade 4 | 0 | 1 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs included body temperature, systolic and diastolic blood pressure, pulse rate, respiratory rate, weight and height. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in vital signs were reported.
Time Frame: up to Week 16
Population: The SAF included all participants who received at least 1 dose of IMP (M2951 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 97 | 98 | 96 | 99
Participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Parameters
Description: Laboratory investigation included hematology, biochemistry, urinalysis and coagulation. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in laboratory parameters were reported.
Time Frame: up to Week 16
Population: The SAF included all participants who received at least 1 dose of IMP (M2951 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 97 | 98 | 96 | 99
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in 12-Lead Electrocardiogram (ECG) Findings
Description: 12-lead ECG recordings included rhythm, heart rate (as measured by RR interval), PR interval, QRS duration, and QT interval. The corrected QT interval (QTcF) was calculated using Fridericia's formula. 12-lead ECG recordings were obtained after the participants have rested for at least 10 minutes in semisupine position. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in 12-lead ECG findings were reported.
Time Frame: up to Week 16
Population: The SAF included all participants who received at least 1 dose of IMP (M2951 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 97 | 98 | 96 | 99
Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Serum Immunoglobulin (Ig) Levels (IgG, IgA, IgM) at Week 2, 4, 8, 12 and 16
Description: Change in the serum levels of IgG, IgA, IgM were assessed.
Time Frame: Baseline, Week 2, 4, 8, 12 and 16
Population: The SAF included all participants who received at least 1 dose of IMP (M2951 or placebo). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signified those participants who were evaluable for the specified category at given time points.
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 95 | 96 | 95 | 99
gram per liter (g/L)
  IgG: Week 2 | -0.02 (1.083) | -0.07 (1.042) | -0.21 (0.968) | -0.09 (1.062)
  IgG: Week 4: number analyzed (Participants) | 94 | 94 | 93 | 96
  IgG: Week 4 | -0.05 (1.465) | -0.15 (1.576) | -0.34 (1.254) | -0.17 (1.168)
  IgG: Week 8: number analyzed (Participants) | 90 | 94 | 87 | 95
  IgG: Week 8 | 0.12 (1.513) | -0.28 (2.052) | -0.37 (1.565) | -0.35 (2.037)
  IgG: Week 12: number analyzed (Participants) | 83 | 89 | 81 | 88
  IgG: Week 12 | 0.47 (1.617) | -0.17 (2.080) | -0.33 (1.493) | -0.23 (1.781)
  IgG: Week 16: number analyzed (Participants) | 60 | 60 | 63 | 67
  IgG: Week 16 | 0.08 (1.829) | -0.14 (2.349) | -0.14 (1.808) | 0.06 (1.960)
  IgA: Week 2 | -0.01 (0.253) | -0.15 (1.187) | 0.00 (0.242) | 0.03 (0.369)
  IgA: Week 4: number analyzed (Participants) | 94 | 94 | 93 | 96
  IgA: Week 4 | -0.05 (0.326) | -0.01 (0.359) | -0.05 (0.333) | 0.02 (0.396)
  IgA: Week 8: number analyzed (Participants) | 90 | 94 | 87 | 95
  IgA: Week 8 | -0.02 (0.346) | -0.16 (1.322) | -0.06 (0.373) | 0.07 (0.567)
  IgA: Week 12: number analyzed (Participants) | 83 | 89 | 81 | 88
  IgA: Week 12 | 0.02 (0.373) | 0.01 (0.444) | -0.08 (0.388) | 0.05 (0.545)
  IgA: Week 16: number analyzed (Participants) | 60 | 60 | 63 | 67
  IgA: Week 16 | 0.01 (0.466) | 0.07 (0.465) | -0.11 (0.380) | 0.05 (0.478)
  IgM: Week 2 | -0.04 (0.198) | -0.04 (0.183) | -0.03 (0.281) | -0.01 (0.323)
  IgM: Week 4: number analyzed (Participants) | 94 | 94 | 93 | 96
  IgM: Week 4 | -0.04 (0.199) | -0.11 (0.224) | -0.11 (0.217) | -0.05 (0.385)
  IgM: Week 8: number analyzed (Participants) | 90 | 94 | 87 | 95
  IgM: Week 8 | -0.03 (0.310) | -0.20 (0.243) | -0.23 (0.327) | -0.10 (0.485)
  IgM: Week 12: number analyzed (Participants) | 83 | 89 | 81 | 88
  IgM: Week 12 | -0.01 (0.265) | -0.20 (0.309) | -0.25 (0.296) | -0.17 (0.406)
  IgM: Week 16: number analyzed (Participants) | 60 | 60 | 63 | 67
  IgM: Week 16 | -0.16 (0.776) | -0.12 (0.436) | -0.22 (0.246) | -0.12 (0.487)

12. Secondary Outcome: Change From Baseline in B Cell Count at Week 2, 4, 8, 12 and 16
Description: Flow cytometry analysis of lymphocyte populations using four-color fluorescence-activated cell sorting was performed for the analysis of B cell counts.
Time Frame: Baseline, Week 2, 4, 8, 12 and 16
Population: SAF included all participants who received at least 1 dose of IMP (M2951 or placebo). Here, "Overall Number of Participants Analyzed specifies those participants who were evaluable for this outcome measure and "Number Analyzed" signified those participants who were evaluable for the specified category at given time point.
Measure: Mean (Standard Deviation); unit: cells per microliter (cells/microliter)
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 90 | 90 | 92 | 97
cells per microliter (cells/microliter)
  Week 2: number analyzed (Participants) | 87 | 90 | 92 | 97
  Week 2 | -13 (111.0) | 264 (1832.7) | 161 (648.3) | 74 (144.8)
  Week 4: number analyzed (Participants) | 90 | 90 | 91 | 93
  Week 4 | -20 (115.7) | 71 (130.1) | 66 (145.3) | 93 (137.6)
  Week 8: number analyzed (Participants) | 81 | 90 | 82 | 91
  Week 8 | -21 (87.5) | 35 (103.1) | 56 (188.1) | 59 (145.4)
  Week 12: number analyzed (Participants) | 82 | 85 | 77 | 83
  Week 12 | -22 (136.4) | 41 (111.8) | 51 (156.2) | 54 (145.0)
  Week 16: number analyzed (Participants) | 56 | 58 | 60 | 64
  Week 16 | -20 (121.9) | -3 (108.5) | -40 (133.5) | -19 (235.6)

13. Secondary Outcome: Percentage of Participants With Remission Assessed by American College of Rheumatology-European League Against Rheumatism (ACR-EULAR) Boolean at Week 12
Description: ACR-EULAR Boolean remission was when a participant satisfied all of the following: tender joint count, swollen joint count (both based on a 28-joint assessment), C-reactive Protein (in milligrams per deciliter [mg/dL]), and participant's global assessment (visual analog scale [VAS]: 0 centimeter (cm) [very well] to 10 cm [worst], higher scores indicated worse health condition) and all scores were less than or equal to (<=) 1. Percentage of participants with ACR-EULAR Boolean Remission were reported.
Time Frame: Week 12
Population: The mITT analysis set included all randomized participants who received at least one dose of IMP (M2951 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 97 | 98 | 96 | 99
percentage of participants | 0.0 | 0.0 | 1.0 | 3.0
Statistical Analysis 1: Comparison: Placebo vs M2951 25 mg QD; Test type: Superiority; Response rate difference = 0.00, 95% CI 2-sided [-0.04 to 0.04]
Statistical Analysis 2: Comparison: Placebo vs M2951 75 mg QD; Test type: Superiority; Response rate difference = 0.01, 95% CI 2-sided [-0.03 to 0.06]
Statistical Analysis 3: Comparison: Placebo vs M2951 50 mg BID; Test type: Superiority; Response rate difference = 0.03, 95% CI 2-sided [-0.01 to 0.09]

14. Secondary Outcome: Percentage of Participants With Clinical Disease Activity Index (CDAI) Score Less Than or Equal to [=<] 2.8 at Week 12
Description: CDAI: a composite index (without acute-phase reactant) for assessing disease activity. The CDAI was calculated based on following formula: CDAI = 28 joint count for swelling (SJC28) + 28 joint count for tenderness (TJC28) + GH + PhGA where, GH = general health component of the Disease Activity Score [DAS] (i.e., Participant's Global Assessment of Disease Activity, assessed using a scale of 0 to 10 centimeter (cm) Visual Analogue Scale (VAS) where 0 = very well and 10 = very poor activity and PhGA = Physician's Global Assessment of Disease Activity assessed using a scale of 0 to 10 cm VAS, where 0 = very well and 10 = very poor activity. The total CDAI score ranges from 0 to 76, where 0 (none) to 76 (extreme disease activity). CDAI score =< 2.8 indicated clinical remission. Percentage of participants with CDAI score =< 2.8 were reported.
Time Frame: Week 12
Population: The mITT analysis set included all randomized participants who received at least one dose of IMP (M2951 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 97 | 98 | 96 | 99
percentage of participants | 1.0 | 4.1 | 6.3 | 3.0
Statistical Analysis 1: Comparison: Placebo vs M2951 25 mg QD; Test type: Superiority; Response rate difference = 0.03, 95% CI 2-sided [-0.02 to 0.09]
Statistical Analysis 2: Comparison: Placebo vs M2951 75 mg QD; Test type: Superiority; Response rate difference = 0.05, 95% CI 2-sided [-0.00 to 0.12]
Statistical Analysis 3: Comparison: Placebo vs M2951 50 mg BID; Test type: Superiority; Response rate difference = 0.02, 95% CI 2-sided [-0.03 to 0.08]

15. Secondary Outcome: Percentage of Participants With Simplified Disease Activity Index (SDAI) Score Less Than or Equal to [=<] 3.3 at Week 12
Description: SDAI was calculated based on following formula: SDAI = 28 joint count for swelling (SJC28) + 28 joint count for tenderness (TJC28) + GH + PGA + hsCRP where, GH = general health component of the Disease Activity Score [DAS] (i.e., Participant's Global Assessment of Disease Activity, assessed using a scale of 0 to 10 centimeter (cm) Visual Analogue Scale (VAS) where 0 = very well and 10 = very poor activity and PhGA = Physician's Global Assessment of Disease Activity assessed using a scale of 0 to 10 cm VAS, where 0 = very well and 10 = very poor activity. The total SDAI score ranges from 0 to 86, where 0 (none) to 86 (extreme disease activity). SDAI score =< 3.3 indicated clinical remission. Percentage of participants with SDAI score =< 3.3 at Week 12 were reported.
Time Frame: Week 12
Population: The mITT analysis set included all randomized participants who received at least one dose of IMP (M2951 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 97 | 98 | 96 | 99
percentage of participants | 0.0 | 3.1 | 4.2 | 3.0
Statistical Analysis 1: Comparison: Placebo vs M2951 25 mg QD; Test type: Superiority; Response rate difference = 0.03, 95% CI 2-sided [-0.01 to 0.09]
Statistical Analysis 2: Comparison: Placebo vs M2951 75 mg QD; Test type: Superiority; Response rate difference = 0.04, 95% CI 2-sided [0.00 to 0.10]
Statistical Analysis 3: Comparison: Placebo vs M2951 50 mg BID; Test type: Superiority; Response rate difference = 0.03, 95% CI 2-sided [-0.01 to 0.09]

16. Secondary Outcome: Percentage of Participants With Good or Moderate European League Against Rheumatism (EULAR) Responses at Week 12
Description: EULAR Responder index based on 28 joint counts categorizes clinical response based on improvement since baseline in DAS28-CRP. DAS28-CRP scores range from 0-9.4, where lower scores indicated less disease activity. High disease activity: DAS28-CRP >5.1, low disease activity: DAS28-CRP <3.2, and remission: DAS28-CRP <2.6. EULAR DAS28-CRP responder index: good (absolute: <3.2 or >1.2 improvement from baseline), moderate (absolute: 3.2-5.1 or 0.6-1.2 improvement from baseline), or no response (absolute: >5.1 or <0.6 improvement from baseline). Percentage of Participants With Good or Moderate EULAR Responses were reported.
Time Frame: Week 12
Population: The mITT analysis set included all randomized participants who received at least one dose of IMP (M2951 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 97 | 98 | 96 | 99
percentage of participants | 54.6 | 65.3 | 66.7 | 71.7
Statistical Analysis 1: Comparison: Placebo vs M2951 25 mg QD; Test type: Superiority; Response rate difference = 0.11, 95% CI 2-sided [-0.03 to 0.24]
Statistical Analysis 2: Comparison: Placebo vs M2951 75 mg QD; Test type: Superiority; Response rate difference = 0.12, 95% CI 2-sided [-0.02 to 0.25]
Statistical Analysis 3: Comparison: Placebo vs M2951 50 mg BID; Test type: Superiority; Response rate difference = 0.18, 95% CI 2-sided [0.05 to 0.31]

17. Secondary Outcome: American College of Rheumatology (ACR) Hybrid Scores Computed Using High-Sensitivity C-reactive Protein (hsCRP)
Description: The hybrid ACR combines the ACR 20/50/70 response with the mean percent change in all 7 ACR core components, thus providing a percent improvement from baseline on a continuous scale. For each participant, the mean percent improvement from baseline across the 7 ACR core set measures (tender joint count, swollen joint count, Patient's Global Assessment of Disease Activity, Physician's Global Assessment of Disease Activity, disability index of the Health Assessment Questionnaire [HAQ], and C-reactive protein [CRP]) was calculated (a positive change indicated improvement, and the maximum worst change was limited to -100%) and the ACR20, ACR50, and ACR70 response is determined. The hybrid ACR is determined from a reference table taking into account both ACR response and mean percent improvement in the core set measures. Scores can range from -100% (maximal worsening) to 100% (maximal improvement).
Time Frame: Baseline, Week 12
Population: The mITT analysis set included all randomized participants who received at least one dose of IMP (M2951 or placebo). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 96 | 97 | 96 | 98
percent change | 26.51 (25.779) | 34.66 (29.033) | 33.09 (27.724) | 36.99 (26.241)

18. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS) Based on a 28 Joint Count-High-Sensitivity C-reactive Protein (DAS28-hsCRP) at Week 12
Description: DAS28 was a composite score used for measuring disease activity in participants with rheumatoid arthritis. The calculation was based on the tender joint count (out of 28 joints), swollen joint count (out of 28 joints), hsCRP (milligrams per liter [mg/L]) and Participant's Global Assessment of Disease Activity. Total DAS28-hsCRP score ranged from 0 (none) to 9.4 (extreme disease activity). DAS28-hsCRP < 3.2 implied low disease activity and >= 3.2 to <= 5.1 implied moderate disease activity, > 5.1 implied high disease activity. DAS28-hsCRP = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(hsCRP in mg/L +1) + 0.014* Participant's Global Assessment of Disease Activity + 0.96; ln = natural logarithm, sqrt = square root.
Time Frame: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 96 | 97 | 96 | 98
units on a scale | -1.21 (1.048) | -1.45 (1.230) | -1.62 (1.257) | -1.75 (1.229)

19. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 12
Description: The CDAI was a composite index (without acute-phase reactant) for assessing disease activity. The CDAI was calculated based on following formula: CDAI = 28 joint count for swelling (SJC28) + 28 joint count for tenderness (TJC28) + GH + PhGA where, GH = general health component of the DAS (i.e., Participant's Global Assessment of Disease Activity, assessed using a scale of 0 to 10 centimeter (cm) Visual Analogue Scale (VAS) where 0 = very well and 10 = very poor activity and PhGA = Physician's Global Assessment of Disease Activity assessed using a scale of 0 to 10 cm VAS, where 0 = very well and 10 = very poor activity. The total CDAI score ranges from 0 to 76, where 0 (none) to 76 (extreme disease activity).
Time Frame: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 96 | 97 | 96 | 98
units on a scale | -16.9 (13.09) | -18.0 (13.00) | -18.9 (14.33) | -20.3 (13.90)

20. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) at Week 12
Description: SDAI was numerical sum of 5 outcome parameters: 28 joint count for swelling (SJC28) + 28 joint count for tenderness (TJC28) + GH + PGA + hsCRP where, GH = general health component of the DAS (i.e., Participant's Global Assessment of Disease Activity, assessed using a scale of 0 to 10 centimeter (cm) Visual Analogue Scale (VAS) where 0 = very well and 10 = very poor activity and PhGA = Physician's Global Assessment of Disease Activity assessed using a scale of 0 to 10 cm VAS, where 0 = very well and 10 = very poor activity. The total SDAI score ranges from 0 to 86, where 0 (none) to 86 (extreme disease activity).
Time Frame: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 96 | 97 | 96 | 98
units on a scale | -17.000 (13.5175) | -18.647 (13.5957) | -19.404 (14.1591) | -21.053 (14.3720)

21. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC) and Swollen Joint Count (SJC) at Week 12
Description: Sixty-eight joints were assessed and classified as tender/not tender and Sixty-six joints were classified as swollen/not swollen by pressure and joint manipulation on physical examination.
Time Frame: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 96 | 97 | 96 | 98
joints
  TJC | -11 (12.0) | -11 (10.6) | -13 (13.2) | -12 (10.8)
  SJC | -7 (7.5) | -8 (6.1) | -8 (7.7) | -8 (6.6)

22. Secondary Outcome: Change From Baseline in Participant's Global Assessment of Disease Activity Based on Visual Analog Scale (VAS) Score at Week 12
Description: The participant's overall assessment of disease activity was recorded using the 100 millimeter (mm) horizontal visual analog scale (VAS). The scale ranged from 0-100 mm, where 0 indicated no disease activity (symptom free and no arthritis symptoms) and 100 represented maximum disease activity (maximum arthritis disease activity).
Time Frame: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 96 | 97 | 96 | 98
millimeter (mm) | -20 (29.6) | -19 (27.9) | -17 (29.6) | -25 (25.7)

23. Secondary Outcome: Change From Baseline in Participant's Assessment of Pain Based on Visual Analog Scale (VAS) Score at Week 12
Description: The participants were asked to assess their level of pain by marking a vertical tick on a 100 mm horizontal VAS scale. The scale ranged from 0-100 mm, where 0 indicated no pain and 100 indicated worst possible pain.
Time Frame: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 96 | 97 | 95 | 98
millimeter | -21 (24.7) | -24 (26.9) | -22 (24.7) | -25 (26.6)

24. Secondary Outcome: Changes From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Total Score at Week 12
Description: HAQ-DI score was an evaluation of the functional status for a participant. The 20-question instrument assessed the degree of difficulty a person had in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0, indicated no difficulty, to 3, indicated inability to perform a task in that area. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range: 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 96 | 97 | 95 | 98
units on a scale | -0.38 (0.567) | -0.58 (0.662) | -0.40 (0.658) | -0.52 (0.616)

25. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity Scale Based on Visual Analog Scale (VAS) Score at Week 12
Description: The Physician's Global Assessment of Disease Activity was recorded using the 100 mm horizontal VAS. Physician rated participant's arthritis disease activity on a scale ranged from 0-100 mm, where 0 indicated no disease activity (no arthritis) and 100 represented maximum disease activity (maximum arthritis).
Time Frame: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 96 | 97 | 96 | 98
millimeter | -29 (21.2) | -33 (26.5) | -34 (26.1) | -37 (25.3)

26. Secondary Outcome: Change From Baseline in High-Sensitivity C-reactive Protein (hsCRP) at Week 12
Description: hsCRP was the American College of Rheumatology (ACR) Core Set measure of acute phase reactant. It was measured at the central laboratory to help assess the effect of M2951 on the participant's rheumatoid arthritis.
Time Frame: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 96 | 97 | 96 | 99
milligram per liter (mg/L) | -1.11 (25.925) | -6.42 (23.280) | -5.45 (28.807) | -7.69 (23.007)

27. Secondary Outcome: Percent Change From Baseline in Tender Joint Count (TJC) and Swollen Joint Count (SJC) at Week 12
Description: as for outcome 21
Time Frame: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 96 | 97 | 96 | 98
percent change
  TJC | -39 (45.6) | -46 (44.2) | -51 (42.8) | -49 (37.5)
  SJC | -46 (52.7) | -53 (42.6) | -56 (40.3) | -58 (43.8)

28. Secondary Outcome: Percent Change From Baseline in Participant's Global Assessment of Disease Activity Based on Visual Analog Scale (VAS) Score at Week 12
Description: as for outcome 22
Time Frame: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 96 | 96 | 96 | 98
percent change | -13 (111.0) | -21 (69.3) | -13 (65.7) | -33 (35.9)

29. Secondary Outcome: Percent Change From Baseline in Participant's Assessment of Pain Based on Visual Analog Scale (VAS) Score at Week 12
Description: as for outcome 23
Time Frame: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 96 | 97 | 95 | 99
percent change | -23 (65.0) | -32 (38.4) | -29 (40.5) | -32 (48.4)

30. Secondary Outcome: Percent Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Total Score at Week 12
Description: as for outcome 24
Time Frame: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 95 | 97 | 95 | 98
percent change | -20.09 (40.084) | -31.85 (37.124) | -21.27 (44.571) | -27.12 (42.624)

31. Secondary Outcome: Percent Change From Baseline in Physician's Global Assessment of Disease Activity Scale Based on Visual Analog Scale (VAS) Score at Week 12
Description: as for outcome 25
Time Frame: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 96 | 97 | 96 | 98
percent change | -42 (31.4) | -44 (51.9) | -47 (34.9) | -52 (33.5)

32. Secondary Outcome: Percent Change From Baseline in High-Sensitivity C-reactive Protein (hsCRP) at Week 12
Description: as for outcome 26
Time Frame: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 96 | 97 | 96 | 99
percent change | 95.01 (380.161) | 10.93 (167.257) | 182.57 (1775.154) | -13.91 (105.688)

33. Secondary Outcome: Change From Baseline in Synovitis Score According to the Outcomes Measures in Rheumatology Clinical Trials Rheumatoid Arthritis Magnetic Resonance Imaging Scoring System (OMERACT RAMRIS) at Week 12
Description: A total of 8 joints in the hand and wrist were evaluated for RAMRIS synovitis. Individual joint scores were assessed on a scale of 0 (no synovitis) to 3 (67 to 100 percent volume enhancement). The final synovitis score was the sum of the individual joint scores. The total score from 8 joints ranges from 0 to 24, with 0 implying normal (no synovitis) and 24 implying 67 to 100 percent volume enhancement.
Time Frame: Baseline, Week 12
Population: The Magnetic Resonance Imaging (MRI) analysis set included all randomized participants who have at least at least 1 pre-dose and 1 post-dose MRI assessment. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 44 | 49 | 47 | 51
units on a scale | 0 (1.9) | -1 (2.5) | -1 (3.4) | -1 (2.4)

34. Secondary Outcome: Change From Baseline in Bone Marrow Edema (Osteitis) Score According to the Outcomes Measures in Rheumatology Clinical Trials Rheumatoid Arthritis Magnetic Resonance Imaging Scoring System (OMERACT RAMRIS) at Week 12
Description: A total of 25 locations in the hand and wrist were evaluated for RAMRIS bone edema or osteitis. Individual location scores range from 0 (no edema) to 3 (67 to 100 percent involvement of original articular bone) based on the proportion of estimated originally non-eroded bone involved. The final bone edema or osteitis score is the sum of the individual location scores. The total score from the 25 locations ranges from 0 to 75, with 0 implying no bone edema or osteitis and 75 implying 67 to 100 percent involvement of original articular bone.
Time Frame: Baseline, Week 12
Population: The MRI analysis set included all randomized participants who have at least at least 1 pre-dose and 1 post-dose MRI assessment. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 44 | 49 | 47 | 51
units on a scale | -1 (5.8) | 0 (4.6) | 0 (5.4) | 0 (4.0)

35. Secondary Outcome: Change From Baseline in Physical Function Using Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 12
Description: The HAQ-DI questionnaire assessed the participant's self-perception on the degree of difficulty [0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do)] when dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities. Scores for each functional area were averaged to calculate HAQ-DI scores, which ranged from 0 (no disability) to 3 (worst disability). A decrease in HAQ-DI score indicated an improvement in the participant's condition.
Time Frame: Baseline, Week 12
Population: Quality of Life (QoL) Analysis Set: all randomized participants who have received at least 1 dose of IMP (M2951 or placebo) and had at least 1 Baseline and 1 post baseline QoL assessment. "Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 87 | 93 | 86 | 92
units on a scale | -0.41 (0.543) | -0.61 (0.637) | -0.45 (0.657) | -0.53 (0.631)

36. Secondary Outcome: Change From Baseline in the Short-Form (SF-36) Health Survey Physical Component Score and Mental Component Score at Week 12
Description: The 36-Item Short-Form Health Survey (SF-36) was a standardized survey evaluating 8 aspects of functional health and well-being. These eight subscales were summarized as relating to either physical health or mental health. Physical component summary (PCS) was based primarily on physical functioning, role-physical, bodily pain, and general health scales and mental component summary (MCS) encompasses vitality, social functioning, role-emotional, and mental health scales. Score from mental health, role emotional, social functioning, and vitality domains were averaged to calculate MCS. Total score range for MCS was 0-100 (100 = highest level of mental functioning). Score from physical function, role physical, bodily pain, and general health domains were averaged to calculate PCS. Total score range for PCS was 0-100 (100 = highest level of physical functioning).
Time Frame: Baseline, Week 12
Population: QoL analysis set: all randomized participants who have received at least 1 dose of IMP (M2951 or placebo) and had at least 1 Baseline and 1 post baseline QoL assessment. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 87 | 93 | 86 | 92
units on a scale
  PCS | 5.9 (7.10) | 7.1 (8.50) | 6.4 (8.50) | 7.1 (8.28)
  MCS | 4.9 (11.46) | 5.7 (8.41) | 5.0 (11.72) | 4.7 (8.95)

37. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Week 12
Description: The FACIT-Fatigue score was calculated according to a 13-item questionnaire that assess self-reported fatigue and its impact upon daily activities and function. It uses a 5-point Likert-type scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; 4 = very much). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse possible score) to 52 (best score). A higher score reflected an improvement in the participant's health status.
Time Frame: Baseline, Week 12
Population: QoL analysis set included all randomized participants who have received at least 1 dose of IMP (M2951 or placebo) and had at least 1 Baseline and 1 post Baseline QoL assessment. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
Number analyzed (Participants) | 87 | 93 | 86 | 92
units on a scale | 9 (11.4) | 10 (9.4) | 9 (9.0) | 8 (10.7)

ADVERSE EVENTS:
Time Frame: up to Week 16
Arm/Group | Placebo | M2951 25 mg QD | M2951 75 mg QD | M2951 50 mg BID
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/98 | 0/96 | 0/99
Serious Adverse Events (participants affected / at risk) | 2/97 | 2/98 | 2/96 | 1/99
Other Adverse Events (participants affected / at risk) | 11/97 | 13/98 | 8/96 | 17/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=97) | M2951 25 mg QD (N=98) | M2951 75 mg QD (N=96) | M2951 50 mg BID (N=99)
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=97) | M2951 25 mg QD (N=98) | M2951 75 mg QD (N=96) | M2951 50 mg BID (N=99)
Anaemia (Blood and lymphatic system disorders) | 6 | 2 | 3 | 7
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 5 | 0 | 2
Headache (Nervous system disorders) | 5 | 6 | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT03233230/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT03233230/SAP_001.pdf